CLINICAL TRIAL: NCT04208074
Title: Enhancing Muscle Strength and Immunity in Breast Cancer
Brief Title: Exercise Study for Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: San Diego Biomedical Research Institute (Other)
Collaborators: California Breast Cancer Research Program (Other); Arizona State University (Other); Tri-City Wellness & Fitness Center (Unknown); We Support U (Unknown)
Responsible Party: Principal Investigator, Joanna Davies, President and CEO, Professor, San Diego Biomedical Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25IB-0023
Record Dates: First submitted 2019-12-10; First posted 2019-12-23 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: Exercise; Resistance Exercise; T cells; Immune system
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Four months of muscle resistance training (exercise) designed to increase muscle mass and strength. The exercise protocol includes four different lifts with weights including, squats, bench press, dead lift and overhead press. The weights for each lift will be optimized for each participant and increased as the participant adapts to the exercise routine.
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — Participants will exercise under the supervision of expert personal trainers and follow an optimized exercise program tailored to the strength and fitness level of each participant. Participants will exercise for 16 weeks; 2 days a week at the gym for an hour and 2 days of the week at home for 45 minutes.

SUMMARY:
This study evaluates the link between muscle health and immune health in breast cancer survivors. Regular exercise is known to improve overall survival in cancer patients but the mechanism is not known. In this study the investigators will evaluate if improving muscle mass and strength via exercise improves the immune system's ability to fight cancer.

This is a one armed study where in 30 breast cancer survivors will be recruited to a 4 month exercise intervention. Increase in muscle mass and strength will be correlated with immune cell frequency and function.

DETAILED DESCRIPTION:
Breast cancer survivors with stronger and larger muscles have better overall survival and lower recurrence than women with weaker and smaller muscles. However, the mechanism for this association is currently unknown. A recent study from the investigators has shown that there is an association between the frequency of immune cell types that kill cancer and higher muscle mass and strength, with higher muscle mass and strength correlating with a higher frequency of cancer killing, effector memory, T cells. The investigators thus propose that increasing muscle mass and strength can improve overall survival and reduce recurrence by increasing the number of cancer killing immune T cells.

To test this hypothesis, the investigators will recruit 30 breast cancer survivors to an exercise program designed to increase their muscle mass and strength. The program will be optimized to each participant's level of fitness and strength and will be designed by experts in the field. Personal trainers will teach the participants how to exercise and use muscle resistance training equipment using the correct technique and will monitor progress to avoid injuries and to maximize training benefits.

The investigators will collect blood (to study immune cell subsets) and measure muscle strength and body composition (to measure muscle mass) for participants before and after the study.

The duration of the exercise training protocol is 4 months and participants will be asked to exercise 4 days a week; 2 days at the gym and 2 days at home.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Post menopausal
* Stage I - III breast cancer
* Breast cancer the only cancer
* Can exercise for 16 weeks; 2 days a week at the gym and 2 days of the week at home
* Live in the San Diego area

Exclusion Criteria:

* Exercise regularly in the gym.
* Are on chemotherapy or radiation therapy or have been in the past month
* Will be on chemotherapy or radiation therapy in the next 6 months
* Have a condition that will prevent them from exercising in the gym

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Since very few men are diagnosed with breast cancer study, women previously diagnosed with breast cancer will be the only group eligible.
Enrollment: 30 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of effector memory immune cells | 16 weeks of muscle resistance training
  Effector memory cells are immune cells that can kill cancer. We will measure the frequency of these cells before and after the 16 week training program to see if they increase. Flow Cytometry techniques will be used to determine the frequency of these cells.
Change in frequency of central memory immune cells | 16 weeks of muscle resistance training
  Central memory cells are immune cells that are linked to poor prognosis in patients with cancer. We will measure the frequency of these cells before and after the 16 week training program to see if they decrease. Flow Cytometry techniques will be used to determine the frequency of these cells.
Change in frequency of regulatory immune cells | 16 weeks of muscle resistance training
  Regulatory immune cells, also called Tregs, are a type of immune cell that keeps the immune system from becoming over active. However, people with too many Treg cells might be more susceptible to cancer growth. We will measure the frequency of Tregs by Flow Cytometry before and after the 16 week training program to see if exercise reduces their frequency.
Change muscle mass | 16 weeks of muscle resistance training
  Dual energy x-ray absorptiometry (DEXA) scans will be used to measure the appendicular muscle mass (amount of muscle in the arms and legs) before and after the 16 week training program. The appendicular muscle mass index is calculated using the appendicular muscle mass divided by height square and is measured in kg/m^2.
Change in hand grip strength | 16 weeks of muscle resistance training
  The level of hand grip strength is a good indicator of body strength. Hand grip strength will be measured in kilograms using an instrument called a dynamometer before and after the 16 week training program.
Change in capacity to climb stairs | 16 weeks of muscle resistance training
  The stair climb test measures the amount of power used by a participant to climb a set of stairs. Power is measured in Watts (W) and is calculated using the time taken to climb the stairs (seconds), the vertical height of the stairs (meters) and the weight (kilograms) of the participant and is a standard measure of performance. The stair climb test will be performed before and after the 16 week training program.
Change in upper body strength | 16 weeks of muscle resistance training
  The Chest Press Test will be used to measure upper body strength. It will be performed before and after the 16 week training program using specialized exercise equipment in the gym. This test will measure the maximum weight that be lifted by the arms and will be measured in kilograms.
Change in lower body strength | 16 weeks of muscle resistance training
  The Knee Extension Test will be used as a measure of lower body strength. It will be performed before and after the 16 week training program using specialized exercise equipment in the gym. This test will measure the maximum weight that be lifted by the legs and will be measured in kilograms.
Change in levels of inflammatory factors in the blood | 16 weeks of muscle resistance training
  The investigators will measure the levels of inflammatory and anti-inflammatory factors, called cytokines, in blood collected before and after the 16 week training program. Cytokines will be measured in picograms per milliliter.
Change in levels of factors called microRNAs in the blood | 16 weeks of muscle resistance training
  The investigators will measure levels of microRNAs in the blood before and after the 16 week training protocol. The microRNAs will be detected and levels measured using a technique called qPCR.

SECONDARY OUTCOMES:
Body Mass Index | 1 day before, and 1 day after the 16 week muscle resistance training program
  BMI will be calculated using height and weight measurements and reported as kg/m2
Physical activity | 1 day before, and 1 day after the 16 week muscle resistance training program
  Physical activity will be determined using the Framingham Physical activity questionnaire. Overall physical activity will be calculated using the physical index score, with a higher score indicating higher physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna D Davies, PhD, Principal Investigator — San Diego Biomedical Research Institute
Locations (1):
- Aditi Narsale, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Narsale A, Moya R, Ma J, Anderson LJ, Wu D, Garcia JM, Davies JD. Cancer-driven changes link T cell frequency to muscle strength in people with cancer: a pilot study. J Cachexia Sarcopenia Muscle. 2019 Aug;10(4):827-843. doi: 10.1002/jcsm.12424. Epub 2019 Apr 12. PMID 30977974
- See also: Information about the study on the official San Diego Biomedical Research Institute website — https://sdbri.org/news-entry/breast-cancer-recruitment/
- See also: Visit us at the link above for more information about the study — https://finance725.wixsite.com/sdbribreastcancer